CLINICAL TRIAL: NCT04424992
Title: Observational Cohort Study on the Natural History of Hospitalized SARS-COV-2 Patients: the STORM Trial
Brief Title: The Natural History of Hospitalized COVID-19 Patients
Acronym: STORM
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: STORM
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Sars-CoV2
Keywords: Coronavirus; sars-covid-2; coronavirus infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum from COVID+ patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Covid19 infection related patients: The patients enrolled in the study are all patients with clinical and microbiological diagnosis of COVID-19 infection hospitalized since February 23, 2020 at San Gerardo Hospital (ASST-Monza).
  Interventions: Other: Observational cohort study on the natural history of hospitalized SARS-COV-2 patients.

INTERVENTIONS:
Other: Observational cohort study on the natural history of hospitalized SARS-COV-2 patients. — Describe the natural history and clinical evolution of hospitalized patients over time affected by SARS-COV-2 infection, understand the pathogenesis of the disease and improve the aids and therapeutic procedures.

SUMMARY:
This is an observational study. The aim is to describe the natural history and clinical evolution over time of hospitalized patients affected by Severe Acute Respiratory Syndrome-Coronavirus-2 (SARS-COV-2) infection, including the genetic pathology of the disease and improve therapeutic procedures.

DETAILED DESCRIPTION:
BACKGROUND:

As of the end of February 2020, the ASST of Monza, with its two hospital wards of Monza and Desio, has treated 1433 COVID+ patients, of which 507 have currently been discharged (35.4%) and 206 (14%) transferred to other Low-intensity care facilities.

The importance of observational studies is now known in many fields of medicine and the "real life" data produced have become an integral part of the authorization dossiers by the competent authorities to govern the introduction of new drugs: in particular, in a disease such as that from COVID-19 in which the absence of specific anti-viral therapies prevents an "ad hoc" cure, it becomes fundamental to identify and validate systems of stratification of the risk of fatal events, in order to optimize health intervention measures.

METHODS AND STUDY DESIGN:

The study protocol provides the collection of clinical, diagnostic and therapeutic and laboratory data consistent with the objectives of the study (CORE DATA SET) to which other specific protocols and relative data will connect (DATABASE "leaf"). The data collection will be performed on eCRF (RedCap platform) and the database will have the "stem and leaf" structure, compatible with WHO indications regarding pandemic data collection.

CORE DATA SET:

The protocol presents two important aspects of innovation in its formulation and design:

1. The "stem and leaf" structure will allow to collect all the core data of the study ("stem") capable of describing the primary objective, that is the natural history of the disease, thus providing an important contribution to knowledge, currently very scarce , the evolution of the disease;
2. the extreme heterogeneity of the pathology itself, the methods of spreading the contagion and the problematic treatment of some particular patient populations, however impose the description and the potential validation, not only in the context of subgroup analyzes, but in studies dedicated, of the data collected The "stem and leaf" design could therefore answer both questions.

BIOLOGICAL SAMPLE COLLECTION:

The biological research areas that the protocol proposes to pursue are listed below:

1. Study of genetic determinants of COVID-19 infection with the aim of identifying the bases of the different susceptibility in relation to age, sex and presence of co-morbidity;
2. Study of the repertoire of B and T lymphocyte receptors and identification of the virus-specific sequences of the T receptor for the antigen with the aim of identifying the component of the viral genome relevant to the immune response with possible relapses for the development of a vaccine;
3. Study of the activation of the inflammosome responsible for the abnormal and severe inflammatory response characteristic of patients with COVID-19 infection and serious lung complications with the aim of identifying possible specific targets of intervention against one or more inflammatory cytokines;
4. Study of the serological response during the acute phase of the disease and convalescence with the aim of defining the possible state of protection from the disease itself;
5. Study of the proteome with the aim of defining biomarkers capable of evaluate the risk of progression.

STATISTICAL ANALYSIS:

For each specific protocol, the study design and statistical data analysis plan will be formulated according to the specific objectives. In general, in addition to the descriptive methods, statistical regression models and methods for the definition of prognostic scores will be used, with relative cross-validation, which will allow to evaluate both binary and survival outcomes (in a broad sense, of events considered in time).

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and / or radiological diagnosis of lung infection with COVID-19;
2. Positive test for SARS-CoV-2 infection.

Exclusion Criteria:

1. Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients enrolled in the study are all patients with clinical and microbiological diagnosis of COVID-19 infection hospitalized since February 23, 2020 at San Gerardo Hospital (ASST-Monza).
Sampling Method: Non-Probability Sample
Enrollment: 1433 (Estimated)
Dates: Start 2020-02-28 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Covid19 infection clinical evolution | Until patient discharge from the hospital (approximately 1 year)
  Description over time of hospitalized patients suffering from SARS-COV-2 infection to better understand the pathogenesis of the disease and improve the controls and therapeutic procedures.

SECONDARY OUTCOMES:
Risk factors for intra-hospital mortality | Until patient discharge from the hospital (approximately 1 year)
  Identify risk factors for intra-hospital mortality in hospital wards COVID + patients.
The impact of a fragility index (IF) | Until patient discharge from the hospital (approximately 1 year)
  Assess the impact of a fragility index (IF) on the clinical course of COVID + patients.
Prognostic score | Until patient discharge from the hospital (approximately 1 year).
  Build a prognostic score through which it is possible define a stratification that orients, according to the state of hospitalization, the therapeutic choices.
The lung sequelae of SARS-COV-2 pneumonia | Until patient discharge from the hospital (approximately 1 year)
  Differentiate the lung sequelae related to the evolution of viral damage from those of cheater / volutrauma connected to non-invasive (NIV-CPAP) or invasive (MV) ventilation methods.
The accuracy of IF in elderly patients | Until patient discharge from the hospital (approximately 1 year)
  Assess the accuracy of IF in elderly patients in terms of clinical outcomes compared to one clinical evaluation based on age and co-morbidity.
Coagulation system anomalies | Until patient discharge from the hospital (approximately 1 year)
  Describe the anomalies of the coagulation system, which appear on patients affected by SARS-COV-2 pneumonia.
The impact of the prone position on the oxygenation | Until patient discharge from the hospital (approximately 1 year)
  Description of the impact of the prone position in terms of increased oxygenation of the patient suffering from SARS-COV-2 pneumonia as an index lung recruitment.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Monza-Ospedale San Gerardo, Monza, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Onder G, Rezza G, Brusaferro S. Case-Fatality Rate and Characteristics of Patients Dying in Relation to COVID-19 in Italy. JAMA. 2020 May 12;323(18):1775-1776. doi: 10.1001/jama.2020.4683. No abstract available. PMID 32203977
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Friesecke S, Stecher SS, Gross S, Felix SB, Nierhaus A. Extracorporeal cytokine elimination as rescue therapy in refractory septic shock: a prospective single-center study. J Artif Organs. 2017 Sep;20(3):252-259. doi: 10.1007/s10047-017-0967-4. Epub 2017 Jun 6. PMID 28589286
- [Background] Yuan FF, Tanner J, Chan PK, Biffin S, Dyer WB, Geczy AF, Tang JW, Hui DS, Sung JJ, Sullivan JS. Influence of FcgammaRIIA and MBL polymorphisms on severe acute respiratory syndrome. Tissue Antigens. 2005 Oct;66(4):291-6. doi: 10.1111/j.1399-0039.2005.00476.x. PMID 16185324
- [Derived] Squillace N, Cogliandro V, Rossi E, Bellelli G, Pozzi M, Luppi F, Lettino M, Strepparava MG, Ferrarese C, Pollastri E, Ricci E, Bonfanti P; STORM Long-COVID Team. A multidisciplinary approach to screen the post-COVID-19 conditions. BMC Infect Dis. 2023 Jan 24;23(1):54. doi: 10.1186/s12879-023-08006-4. PMID 36694110
- [Derived] Coppadoro A, Benini A, Fruscio R, Verga L, Mazzola P, Bellelli G, Carbone M, Mulinacci G, Soria A, Noe B, Beck E, Di Sciacca R, Ippolito D, Citerio G, Valsecchi MG, Biondi A, Pesci A, Bonfanti P, Gaudesi D, Bellani G, Foti G. Helmet CPAP to treat hypoxic pneumonia outside the ICU: an observational study during the COVID-19 outbreak. Crit Care. 2021 Feb 24;25(1):80. doi: 10.1186/s13054-021-03502-y. PMID 33627169